CLINICAL TRIAL: NCT06535009
Title: A Phase I, Open-label, Uncontrolled, Dose Escalation Study to Evaluate the Tolerability and Safety of ONO-7914 Alone and in Combination With ONO-4538 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study of ONO-7914 Alone and in Combination With ONO-4538 in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to strategic reasons
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7914-01
Record Dates: First submitted 2024-07-21; First posted 2024-08-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-7914 (Experimental)
  Interventions: Drug: ONO-7914
- ONO-7914+ONO-4538 (Experimental)
  Interventions: Drug: ONO-7914; Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-7914 — Specified dose on specified days
Drug: ONO-4538 — Specified dose on specified days
  Arms: ONO-7914+ONO-4538

SUMMARY:
This study is dose escalation study to evaluate the tolerability and safety of ONO-7914 alone and in combination with ONO-4538 in patients with advanced or metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic solid tumor
2. Patients with ECOG performance status of 0 or 1
3. Patients with a life expectancy of at least 3 months

Exclusion Criteria:

1. Patients with severe complication
2. Patients judged to be incapable of providing consent for reasons such as concurrent dementia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 days
Adverse Events as assessed by CTCAE v5.0 | Up to 28 days after the completion of treatment period

SECONDARY OUTCOMES:
Plasma concentration of ONO-7914 | Up to 21 days after the first treatment
Urine concentration of ONO-7914 | Up to 24 hours after the first treatment
Serum concentration of ONO-4538 | Up to 28 days after the completion of treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Cancer Institute Hospital of JFCR, Koto-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No